CLINICAL TRIAL: NCT00214123
Title: The Use of Helical Tomotherapy to Achieve Dose-per-fraction Escalation in Lung Cancer
Brief Title: Hypofractionated Radiotherapy for Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RO04502; A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison); NCI-2011-00868 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Bin 1 (Experimental): bin assignment based on tumor volume
  Interventions: Radiation: radiation therapy (radiotherapy)
- Bin 2 (Experimental): Bin assignment based on tumor volume
  Interventions: Radiation: radiation therapy (radiotherapy)
- Bin 3 (Experimental): Bin assignment based on tumor volume
  Interventions: Radiation: radiation therapy (radiotherapy)
- Bin 4 (Experimental): Bin assignment based on tumor volume
  Interventions: Radiation: radiation therapy (radiotherapy)
- Bin 5 (Experimental): Bin assignment based on tumor volume
  Interventions: Radiation: radiation therapy (radiotherapy)

INTERVENTIONS:
Radiation: radiation therapy (radiotherapy) — Bin assignment based on tumor volume

SUMMARY:
The purpose of this trial is to pilot reducing the duration of radiation treatment for lung cancer patients from 6 to 5 weeks using tomotherapy. Specific patient doses will be based on tumor volume being treated. Modeling has shown that increased biologically effective dose (BED) to tumors can be achieved by shortening the radiation delivery schedule and increasing the dose per fraction. This requires decreasing the total dose to hold lung toxicity constant at each dose per fraction level. This is a major paradigm shift in the treatment in this disease and is projected to result in significant improvements in patient outcome as well as a substantial cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic neoplasm requiring at lest 60 Gy conventional radiotherapy

Exclusion Criteria:

* Prior bleomycin or gemcitabine chemotherapy
* Prior thoracic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Grade 3 pneumonitis lasting greater than 2 weeks | 90 days post radiotherapy (XRT)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Cannon DM, Mehta MP, Adkison JB, Khuntia D, Traynor AM, Tome WA, Chappell RJ, Tolakanahalli R, Mohindra P, Bentzen SM, Cannon GM. Dose-limiting toxicity after hypofractionated dose-escalated radiotherapy in non-small-cell lung cancer. J Clin Oncol. 2013 Dec 1;31(34):4343-8. doi: 10.1200/JCO.2013.51.5353. Epub 2013 Oct 21. PMID 24145340